CLINICAL TRIAL: NCT06067438
Title: A Prospective, Randomized Controlled Trial Evaluating the Efficacy of Amiodarone in the Prevention of Postoperative Atrial Fibrillation in Patients Undergoing Minimally Invasive Esophagectomy
Brief Title: Amiodarone for the Prevention of Atrial Fibrillation After Minimally Invasive Esophagectomy in Patients With Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Stephanie Wood, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00021572; NCI-2023-03642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021572 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-06-01; First posted 2023-10-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Esophageal Carcinoma
MeSH Terms: conditions — Atrial Fibrillation; Esophageal Neoplasms | interventions — Amiodarone; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (amiodarone hydrochloride) (Experimental): Patients receive amiodarone hydrochloride IV for 4 days and then via a feeding tube for 3 days on study.
  Interventions: Drug: Amiodarone Hydrochloride
- Arm II (normal saline) (Placebo Comparator): Patients receive normal saline IV for 4 days on study.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Amiodarone Hydrochloride — Given IV and via feeding tube
  Other Names: Cordarone; Nexterone
  Arms: Arm I (amiodarone hydrochloride)
Other: Saline — Given IV
  Other Names: ISOTONIC SODIUM CHLORIDE SOLUTION; Sodium Chloride 0.9%
  Arms: Arm II (normal saline)

SUMMARY:
This phase II trial studies how well amiodarone works in the prevention of atrial fibrillation (AF) after a minimally invasive esophagectomy (MIE) in patients with esophageal cancer. Atrial fibrillation (AF) is an irregular heart rhythm, usually associated with a rapid rate, that is caused by abnormal electrical activity within the atria. AF is the most common complication after MIE for esophageal cancer. There has never been a study of AF after MIE that has used unbiased assignment of patients to receive preventative amiodarone or not. Further, there is no standard recommendation or guideline for preventative medications, such as amiodarone, to decrease the risk of AF in patients having MIE performed for cancer. In fact, most medical centers in the United States and around the world do not give preventative amiodarone after esophagectomy. Giving amiodarone after MIE surgery may be able to reduce the risk of AF for patients with esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of prophylactic amiodarone on the rate of atrial fibrillation (AF) in patients undergoing minimally invasive esophagectomy (MIE).

SECONDARY OBJECTIVES:

I. In each subobjective, below, evaluations of the effects of prophylactic amiodarone on the following will be made:

* Ia. Postoperative (PostOp) rapid ventricular response;
* Ib. Postop pulmonary complications;
* Ic. Postop anastomotic leak;
* Id. Intensive care unit (ICU) readmission;
* Ie. ICU length of stay (LOS);
* If. Hospital LOS;
* Ig. 30-day readmission;
* Ih. Inpatient mortality;
* Ii. 30-day mortality;
* Ij. Adverse events;
* Ik. Time to AF;

Il. Evaluating the association between therapeutic (or serum levels and the development of AF in the experimental group only.

EXPLORATORY OBJECTIVE:

I. To evaluate the effect of prophylactic amiodarone administration on hospital cost of care.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive amiodarone hydrochloride intravenously (IV) for 4 days and then via a feeding tube for 3 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo (normal saline) IV for 4 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for 60 days following discharge from hospitalization after MIE.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing MIE will be evaluated for potential enrollment

  * Indication of cancer, esophageal dysplasia or esophageal dysmotilities
* Age > 18 years
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of chronic or paroxysmal AF, or atrial flutter
* Previous severe adverse reaction or contraindication to amiodarone (e.g., pulmonary toxicity/fibrosis, hepatotoxicity, thyroid dysfunction)
* Current preoperative use of amiodarone, as baseline home medication
* Development of AF intraoperatively
* Pregnancy

  * Negative pregnancy tests are required for participants of childbearing potential (PCBP) on Day of Surgery (DOS)
* Breastfeeding/chest feeding
* Aborted MIE operation
* QTcF (Fridericia formula) > 500 for heart rate (HR) 60-100 within 30 days

  * For patients with a heart rate (HR) of between 50-59 on their pre-operative screening electrocardiography (EKG), we will first review evidence of chronotropic cardiac response to exercise before inclusion in the study. If a patient's HR increases to ≥ 100 with exercise, the patient is eligible for inclusion of study. Exercise testing options may include a stair climb, a brisk walk, or supine leg-lifts prior to surgery. If exercise is not an option, we can review results of formal stress testing chronotropic response (ie. HR ≥ 100). HR monitoring can be collected by either pulse oximeter or EKG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Development of atrial fibrillation (AF), or completion of seven-day course of amiodarone | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 7, after last dose of enteral amiodarone
  Will be a binary variable (yes/no) and analyzed using a one-sided test of two proportions at an alpha level of 0.05.

SECONDARY OUTCOMES:
Postoperative (PostOp) rapid ventricular response | From initiation of amiodarone in the intensive care unit (ICU) to discharge (DC) from hospital.
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% confidence interval (CI) of the difference between the two proportions.
Postop pulmonary complications | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 30
  Including pneumonia, acute respiratory distress syndrome, acute pulmonary edema, and chylothorax. Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
Anastomotic leak | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 30
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
ICU Readmission | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 30
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
ICU length of stay (LOS) | From initiation of amiodarone in the intensive care unit (ICU) to time patient is moved out of ICU
  Will be assessed in days. Analysis: Wilcoxon rank sum test
Hospital LOS | From initiation of amiodarone in the intensive care unit (ICU) to time of discharge from hospital
  Will be assessed in days. Analysis: Wilcoxon rank sum test
30 Day readmission rate | Day of discharge (DC) from hospital to 30 days after discharge
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
Inpatient morality | From initiation of amiodarone in the intensive care unit (ICU) to time of discharge from hospital
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
Incidence of mortality within 30 days of surgery | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 30
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
Incidence and type of adverse events | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 30
  Will be a binary value (yes/no). Analysis: Binomial test; point estimate and 95% CI of the difference between the two proportions.
Time to AF | From initiation of amiodarone in the intensive care unit (ICU) to post-operative day (POD) 7
  Analysis: Log-rank test.
Serum amiodarone level, classified as therapeutic or subtherapeutic | Post-operative day (POD) 2 to post-operative day (POD) 3

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wood, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided